CLINICAL TRIAL: NCT05187507
Title: The Effectiveness Evaluation of the Theobromine Containing Toothpastes in Controlling Dental Plaque in Children Aged 6-9years(Randomized Controlled Clinical Trial)
Brief Title: Effectiveness of Theobromine Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UDDS-Pedo-06-2021
Record Dates: First submitted 2021-12-24; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Dental Plaque; Dental Care
Keywords: Dental Primary Prevention; Theobromine toothpaste; Fluoridated toothpaste
MeSH Terms: conditions — Dental Plaque | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Children using fluoridated toothpaste (Other)
  Interventions: Other: Evaluation of the effectiveness of fluoridated toothpaste.
- Children using low- fluoridated toothpaste (Other)
  Interventions: Other: Evaluation of the effectiveness of low- fluoridated toothpaste.
- Children using Theobromine toothpaste (2%). (Experimental)
  Interventions: Other: Evaluation of the effectiveness of theobromine toothpaste (2%) toothpaste.
- Children using Theobromine toothpaste(4%) (Experimental)
  Interventions: Other: Evaluation of the effectiveness of theobromine toothpaste(4%) toothpaste.

INTERVENTIONS:
Other: Evaluation of the effectiveness of low- fluoridated toothpaste. — Children will be given low- fluoridated toothpaste, plaque score in groups will be assess pre given toothpaste in baseline,aweek,2week,and after 3weeks by using the TMQHPI for both buccal and lingual surface.
  Gingivalitis will be assess pre given toothpaste,aweek,2weeks,and after 3weeks by using gingival index (loe and silness).
  Arms: Children using low- fluoridated toothpaste
Other: Evaluation of the effectiveness of fluoridated toothpaste. — Children will be given e fluoridated toothpaste, plaque score in groups will be assess pre given toothpaste in baseline,aweek,2week,and after 3weeks by using the TMQHPI for both buccal and lingual surface.
  Gingivalitis will be assess pre given toothpaste,aweek,2weeks,and after 3weeks by using gingival index (loe and silness).
  Arms: Children using fluoridated toothpaste
Other: Evaluation of the effectiveness of theobromine toothpaste (2%) toothpaste. — Children will be given theobromine toothpaste(2%),plaque score in groups will be assess pre given toothpaste in baseline,aweek,2week,and after 3weeks by using the TMQHPI for both buccal and lingual surface.
  Gingivalitis will be assess pre given toothpaste,aweek,2weeks,and after 3weeks by using gingival index (loe and silness).
  Arms: Children using Theobromine toothpaste (2%).
Other: Evaluation of the effectiveness of theobromine toothpaste(4%) toothpaste. — Children will be given theobromine toothpaste(4%),plaque score in groups will be assess pre given toothpaste in baseline,aweek,2week,and after 3weeks by using the TMQHPI for both buccal and lingual surface.
  Gingivalitis will be assess pre given toothpaste,aweek,2weeks,and after 3weeks by using gingival index (loe and silness).
  Arms: Children using Theobromine toothpaste(4%)

SUMMARY:
Since plaque control forms the basis for caries prevention, the type of toothpaste and its constituents becomes more important.

Toothpaste containing fluoride are widely popular and fluorides have been historically reported to have effects against dental caries. However, the fluoride safe doses are still discussed ,because fluoride has toxicity and causing fluorosis.

The aim of the current research is to find alternative agent that can be used without side effects.

DETAILED DESCRIPTION:
Participants will be examined to ensure that they have met the smple entrey criteria,then the participants will be randomly assigned to four groups each one according to a group:

1. A group of children using low-fluoridated toothpaste (500ppm)
2. A group of children using fluoridated toothpaste (1450ppm)
3. A group of children using theobromine toothpaste (2%)
4. A group of children using low-fluoridated toothpaste (4%) The researcher will teach the participants how to brush using (tell-show-do)technique.

   * The brushing method that will be used is the fones technique.
   * Brushing duration must be 2minutes.
   * Frequency of brushing must be twice a day
   * The amount of toothpaste used is pea size.

Mechanism of examination and follow up:

A thorough scaling and plaque removal was conducted and the children were advised to brush their teeth using their regular toothpaste for a week before starting the research.

Gingival will be evaluated with gingival index (loe and silness)

ELIGIBILITY:
Inclusion Criteria:

* Children of age group 6to 9 years.
* Participant must have least 20 teeth free from dental cries on both buccal and lingual surfaces of the teeth.
* Cooperative children having behavioral rating (positive or definitively positive)according to frankel's behavior rating scale.
* Children who are not on any medication prior or during the study period

Exclusion Criteria:

* children with systemic diseases and medically compromising conditions.
* children undergoing orthodontic treatment or with an intraoral prosthesis.
* children who could not brush their teeth or rinse on their own.
* Allergic to any of the toothpaste ingredient used the study.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of using low- fluoridaed toothpaste for children | 1 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using low- fluoridaed toothpaste for children | 2 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using low- fluoridaed toothpaste for children | 3 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using fluoridated toothpaste for children | 1 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using fluoridated toothpaste for children | 2 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using fluoridated toothpaste for children | 3 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using theobromine toothpaste(2%) for children | 1 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using theobromine toothpaste(2%) for children | 2 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using theobromine toothpaste(2%) for children | 3 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using theobromine toothpaste(4%) for children | 1 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using theobromine toothpaste(4%) for children | 2 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).
Clinical evaluation of using theobromine toothpaste(4%) for children | 3 week
  Plaque scores will be assess by using the Turesky Modification of the Quigley-Hein Plaque Index(TMQHPI) for both buccal and lingual surfaces. Plaque will detect using plaque disclosing agent.
  Gingival scores will be assessed with gingival index(loe and silness).

CONTACTS AND LOCATIONS:
Overall Officials: Nour M Zaaweet, DDS, Principal Investigator — MSc student in Pedodontics, University of Damascus; Ettihad A Abo-Arraj, Phd, Study Chair — Professor of Pedodontics, Department of Pedodontics, University of Damascus
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farooq I, Samad Khan A, Moheet IA, Alshwaimi E. Preparation of a toothpaste containing theobromine and fluoridated bioactive glass and its effect on surface micro-hardness and roughness of enamel. Dent Mater J. 2021 Mar 31;40(2):393-398. doi: 10.4012/dmj.2020-078. Epub 2020 Nov 19. PMID 33208577
- [Background] Premnath P, John J, Manchery N, Subbiah GK, Nagappan N, Subramani P. Effectiveness of Theobromine on Enamel Remineralization: A Comparative In-vitro Study. Cureus. 2019 Sep 17;11(9):e5686. doi: 10.7759/cureus.5686. PMID 31720155
- [Background] Lakshmi A, Vishnurekha C, Baghkomeh PN. Effect of theobromine in antimicrobial activity: An in vitro study. Dent Res J (Isfahan). 2019 Mar-Apr;16(2):76-80. PMID 30820200
- [Background] Thorn AK, Lin WS, Levon JA, Morton D, Eckert GJ, Lippert F. The effect of theobromine on the in vitro de- and remineralization of enamel carious lesions. J Dent. 2020;103S:100013. doi: 10.1016/j.jjodo.2020.100013. Epub 2020 Feb 17. PMID 34059300
- [Background] Lippert F. The effects of fluoride, strontium, theobromine and their combinations on caries lesion rehardening and fluoridation. Arch Oral Biol. 2017 Aug;80:217-221. doi: 10.1016/j.archoralbio.2017.04.022. Epub 2017 Apr 20. PMID 28458181